CLINICAL TRIAL: NCT04494880
Title: Marcaine Post-Operative Pain Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1618426-3
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Marcaine 1 Breast) (Experimental): Marcaine will be injected into one randomized breast and saline into the other in the treatment group.
  Interventions: Drug: Bupivacaine Injection
- Control Group (Marcaine 2 Breasts) (No Intervention): Marcaine will be injected into both breasts as is currently the standard of care.

INTERVENTIONS:
Drug: Bupivacaine Injection — Treatment group receives Marcaine (Bupivacaine) injected into one breast following breast reduction surgery and a saline injection in the other group.
  Other Names: Marcaine
  Arms: Treatment Group (Marcaine 1 Breast)

SUMMARY:
The study examines the efficacy of Marcaine in post-operative pain reduction for patients receiving breast reduction surgery. Patients who consent will be randomized to which breast receives a Marcaine injection and the other breast will have saline injected. Pain will be assessed one time post-operatively using a 1-10 pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Must be receiving bilateral breast reduction surgery

Exclusion Criteria:

* Unilateral breast reduction surgery

Max Age: 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Marcaine Use in Breast Reconstruction: Post-Operative Pain Scale Assessment per Breast | through study completion, an average of 1 year
  Minimum score: 1 (minimal pain), Maximum score: 10 (worst pain possible/worst outcome), higher pain scores associated with worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Upadhyaya, MD, Principal Investigator — SUNY Upstate Medical University - Syracuse, NY
Locations (1):
- Upstate University Hospital, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No